CLINICAL TRIAL: NCT00838734
Title: Compare Anterior Chamber Biometry in Healthy and Post-LASIK Pati
Brief Title: Compare Anterior Chamber Biometry in Healthy and Post-LASIK Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Shu-Wen Chang, Far Eastern Memorial Hospital
Other Study IDs: FEMH97011
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Myopia; Astigmatism
Keywords: CORNEAL TOPOGRAPHY; KERATOPLASTY
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Pre-LASIK
- 2: Post-LASIK

SUMMARY:
In this study, the investigators employed Visante-OCT (Carl Zeiss, USA), an anterior chamber optical coherence tomography, to monitor the change of anterior chamber dimensions. These data were correlated to anterior and posterior curvature changes collected with the Oculus Pentacam (Oculus Inc., Germany), a corneal topographer based on rotating Scheimpflug principle. To minimize the effect of convergence and excyclotorsion during examination, topical cycloplegic medication was used. The investigators hypothesized that if there is a link between ciliary muscle contraction and cornea curvature, installation of cycloplegic should result in widening of anterior chamber angle to angle distance and flattening of the cornea curvature data.

DETAILED DESCRIPTION:
Accommodation is an action that enables projections of both distant and near objects to be brought into clear focus on the retina through changing of diopteric power of crystalline lens. Although the exact mechanism of accommodation remains inconclusive, most authors agree that contraction of ciliary muscle plays a pivotal role.1, 2 Recently, accumulating evidence shows that the effect of ciliary muscle contraction goes beyond merely changing the curvature of the crystalline lens.3 Ciliary muscle contraction might be responsible for a transient elongation in axial length during the accommodation response.3 Contraction of ciliary smooth muscle applied an inward pulling force on the choroid and sclera adjacent to the ciliary body and cause protrusion at posterior sclera.

If ciliary muscle contraction can elicit protrusion at posterior sclera, it is conceivable that some changes in corneal shape would also occur as the cornea is adjacent to ciliary muscle. The influence of accommodation on the cornea has therefore been the subject of several studies with conflicting results. Some authors reported no change4, 5, while others described significant change in corneal curvature during accommodation6-9. Yasuda and Yamaguchi9 found central corneal steepening of approximately 0.10 D, using pharmacologically induced ciliary muscle contraction and corneal topography analysis. Saitoh et al10 reported that instillation of a sympathomimetic agent to stimulate mydriasis induces significant flattening of both anterior and posterior cornea curvatures as detected by Orbscan . On the contrary, Buehren5 and Read4 argue that changes in corneal topography is a result of excyclotorsional eye movement during accommodation. When this excyclotorsional eye movement was accounted for in their data analysis, no significant change in corneal topography was found with accommodation. The effect of ciliary relaxation on the cornea curvature, however, was less well delineated.

In this study, we employed Visante-OCT (Carl ZeiIn this study, we employed Visante-OCT (Carl Zeiss, USA), an anterior chamber optical coherence tomography, to monitor the change of anterior chamber dimensions. These data were correlated to anterior and posterior curvature changes collected with the Oculus Pentacam (Oculus Inc., Germany), a corneal topographer based on rotating Scheimpflug principle. To minimize the effect of convergence and excyclotorsion during examination, topical cycloplegic medication was used. We hypothesized that if there is a link between ciliary muscle contraction and cornea curvature, installation of cycloplegic should result in widening of anterior chamber angle to angle distance and flattening of the cornea curvature data.

ss, USA), an anterior chamber optical coherence tomography, to monitor the change of anterior chamber dimensions. These data were correlated to anterior and posterior curvature changes collected with the Oculus Pentacam (Oculus Inc., Germany), a corneal topographer based on rotating Scheimpflug principle. To minimize the effect of convergence and excyclotorsion during examination, topical cycloplegic medication was used. We hypothesized that if there is a link between ciliary muscle contraction and cornea curvature, installation of cycloplegic should result in widening of anterior chamber angle to angle distance and flattening of the cornea curvature data.

In addition, we would also compare the accuracy in pupil diameter measurements between Pentacam and Visante OCT under under normal and mydratic conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy young volunteer who has not received any ocular surgery
* post-LASIK surgery young volunteers
* all participants has to be less than 35 years old.

Exclusion Criteria:

* any subject with contact lens history will be asked to stop contact lens wear for at least 4 weeks before participating in this study.
* any subject with prior ocular disease
* any subject with prior intra-ocular surgery
* any subject who cannot cooperate with examination

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Study Completion 2009-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Wen Chang, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan